CLINICAL TRIAL: NCT00677170
Title: An Open-Label, Dose Escalation, Phase I Study of MLN4924, a Novel Inhibitor of Nedd8-Activating Enzyme, in Adult Patients With Nonhematologic Malignancies
Brief Title: Study of MLN4924 in Adult Patients With Nonhematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C15001
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Advanced Nonhematologic Malignancies
MeSH Terms: interventions — pevonedistat

ARMS (1):
- 1 (Experimental): MLN4924
  Interventions: Drug: MLN4924

INTERVENTIONS:
Drug: MLN4924 — IV dose escalation for 5 consecutive days followed by a rest period of 16 days for a 21 day cycle. Treated may continue until disease progression or unacceptable toxicity develops.

SUMMARY:
This study is an open-label, multicenter, Phase 1, dose escalation study of MLN4924 in adult patients with nonhematologic malignancies. This study will be the first to administer MLN4924 in humans. The patient population will consist of adults with any form of nonhematologic malignancy for which standard, curative, life prolonging, or palliative treatment does not exist or is no longer effective.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Eastern Cooperative Oncology Group performance status 0-2
* Patients must have a diagnosis of a nonhematologic malignancy for which standard curative, life-prolonging, or palliative treatment does not exist or is no longer effective.
* Expected survival longer than 6 weeks from enrollment in the study
* Radiographically or clinically evaluable tumor
* Suitable venous access for the conduct of blood sampling for MLN4924
* Tumor tissue that, in the opinion of the investigator, can be safely biopsied using a core needle
* Male patients must use an appropriate method of barrier contraception
* Female patients must be postmenopausal, surgically sterilized, or willing to use reliable methods of birth control
* Voluntary written consent

Exclusion Criteria:

* Pregnant or lactating
* Major surgery within 14 days prior to the first dose of study treatment
* Serious infection within 14 days prior to the first dose of study treatment
* Receiving antibiotic therapy within 14 days prior to the first dose of study treatment
* Life-threatening illness unrelated to cancer
* Diarrhea that is greater than Grade 1 in severity
* Systemic antineoplastic therapy within 21 days preceding first dose of study treatment
* Radiotherapy within 21 days preceding first dose of study treatment
* Prior treatment with radiation therapy involving ≥25% of the hematopoietically active bone marrow
* CYP3A inducers within 14 days before the first dose of MLN4924. Moderate and strong CYP3A inhibitors and CYP3A inducers are not permitted during the study.
* Clinically significant central nervous system metastases
* Absolute neutrophil count <1,500/mm3; platelet count <100,000/mm3
* Patients with a prothrombin time or aPTT > 1.5 x the upper limit of the normal range, or with a history of a coagulopathy or bleeding disorder
* Ongoing anti-coagulant therapy that can not be held to permit tumor biopsy
* Calculated creatinine clearance <50 mL/minute
* Bilirubin >1.5 times the upper limit of normal; aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase >2.5 times the upper limit of normal.
* Uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months
* Abnormalities on 12-lead electrocardiogram including, but not limited to, changes in rhythm and intervals that in the opinion of the investigator are considered to be clinically significant
* Known human immunodeficiency virus positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Treatment with any investigational products within 28 days preceding the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determine the safety profile, MTD and PK/pharmacodynamics of MLN4924 | Maximum duration of therapy for 12 months

SECONDARY OUTCOMES:
Disease response | Day 21, every other cycle and end of study

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Cancer Therapy & Research Center at the UT Health Science Center, San Antonio, Texas
  - Institute for Drug Development, San Antonio, Texas

REFERENCES:
- [Derived] Faessel HM, Mould DR, Zhou X, Faller DV, Sedarati F, Venkatakrishnan K. Population pharmacokinetics of pevonedistat alone or in combination with standard of care in patients with solid tumours or haematological malignancies. Br J Clin Pharmacol. 2019 Nov;85(11):2568-2579. doi: 10.1111/bcp.14078. Epub 2019 Sep 4. PMID 31355467
- [Derived] Swords RT, Watts J, Erba HP, Altman JK, Maris M, Anwer F, Hua Z, Stein H, Faessel H, Sedarati F, Dezube BJ, Giles FJ, Medeiros BC, DeAngelo DJ. Expanded safety analysis of pevonedistat, a first-in-class NEDD8-activating enzyme inhibitor, in patients with acute myeloid leukemia and myelodysplastic syndromes. Blood Cancer J. 2017 Feb 3;7(2):e520. doi: 10.1038/bcj.2017.1. No abstract available. PMID 28157218